CLINICAL TRIAL: NCT00556816
Title: COPD-C: COPD Outpatient on Demand Clinic. Study to Determine the Efficacy and Safety of on Demand Outpatient Clinics in COPD Patients
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Outpatient on Demand Clinic
Acronym: COPD-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jan W.K. van den Berg, Dr., Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL 14887.075.06
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; outpatient on demand clinic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional outpatient clinic (Active Comparator): Conventional outpatient clinic
  Interventions: Behavioral: Control
- On demand outpatient clinic (Experimental): On demand outpatient clinic
  Interventions: Behavioral: on demand clinic

INTERVENTIONS:
Behavioral: on demand clinic — Outpatient on demand clinic
  Arms: On demand outpatient clinic
Behavioral: Control — conventional outpatient clinic
  Arms: Conventional outpatient clinic

SUMMARY:
COPD (chronic obstructive pulmonary disease) is a chronic disease which is increasing. Patients with COPD are the most important concern of the pulmonologists. At the outpatient clinic has been observed that the amount of new and regular COPD patients is of such a size that it seems to overwhelm the capacity of the outpatient clinic. Solutions could be substitution of medical care, longer intervals between the appointments or discharge from secondary medical care to primary care. The first point does not solve the lack of capacity, the second point is not allowed because it will decrease quality of care and transition of care is a temporary solution. COPD is a complex disease, whereby, and certainly in an advanced stadium, multidisciplinary and qualified expertise is needed.

The optimal control frequency of patients with COPD is unknown. COPD is a disease with fluctuating activity and complaints over time. There is a chance that patients are seen at a stable state at the regular outpatient clinical visits instead of moments when medical care is obligated. The regular management of the outpatient clinic will therefore result in an ineffective treatment of COPD patients. In this way general practitioners and even patients could suggest that visits to the outpatient pulmonary clinic are confounding less to a good treatment of COPD.

Outpatient clinical care on demand, initiated by patients in other chronic patient groups like rheumatoid arthritis and inflammatory bowel diseases, are proven to be safe and effective leading to less consumption and costs of medical care in comparison to standard outpatient clinical visits 2-5.

The outpatient clinical care on demand for COPD is not figured out yet. Our aim is to investigate whether this special type of outpatient clinical care is effective in the management of COPD.

DETAILED DESCRIPTION:
COPD (chronic obstructive pulmonary disease) is a chronic disease with an increasing prevalence in the next years. There has been calculated that between 1994 and 2015 COPD will increase for men and women with 43% and 142%. This will be caused by ageing of the population and the tendency towards more smoking women 1.

Patients with COPD are the most important concern of the pulmonologists. At the outpatient clinic, it has been observed that the amount of new and regular COPD patients is of such a size that it seems to overwhelm the capacity of the outpatient clinic. Solutions could be substitution of medical care (specialist replacement by nurse practitioner), longer intervals between the appointments, or discharge from secondary medical care to primary care. The first point doesn't solve the lack of capacity, the second point is not allowed because it will decrease quality of care, and transition of care is a temporary solution. COPD is a complex disease, whereby, and certainly in an advanced stadium, multidisciplinary and qualified expertise is needed.

The optimal control frequency of patients with COPD is unknown. COPD is a disease with fluctuating activity and complaints over time. There is a chance that patients are seen at a stable state at the regular outpatient clinical visits instead of moments when medical care is obligated. The regular management of the outpatient clinic will therefore result in an ineffective treatment of COPD patients. In this way, general practitioners and even patients could suggest that visits to the outpatient pulmonary clinic are confounding less to a good treatment of COPD.

Outpatient clinical care on demand, initiated by patients in other chronic patient groups like rheumatoid arthritis and inflammatory bowel diseases, are proven to be safe and effective leading to less consumption and costs of medical care in comparison to standard outpatient clinical visits 2-5.

The outpatient clinical care on demand for COPD is not figured out yet. The investigators' aim is to investigate whether this special type of outpatient clinical care is effective in the management of COPD

ELIGIBILITY:
Inclusion Criteria:

* COPD patients at least GOLD II (FEV1 < 70%, FEV1/VC ratio < 70%)
* age > 40 years
* smoking history > 10 pack years
* informed consent

Exclusion Criteria:

* significant or instable comorbidity
* a history of asthma
* drug or alcohol abuse
* incapacity to fill in questionnaires

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
change in health status (CCQ) | 2 years

SECONDARY OUTCOMES:
use of medical care (visits to GP, ER, outpatient clinic) | 2 years
quality of life (SGRQ and SF-36) | 2 years
the number of appointments with the pulmonary nurse/ nurse practitioner | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: L.N. Boom, Drs., Principal Investigator — Isala
Locations (1):
- Isala Klinieken, Zwolle, Netherlands